CLINICAL TRIAL: NCT02908269
Title: Safety and Immunogenicity of Fluzone® Quadrivalent and Fluzone® High-Dose, Influenza Vaccines, 2016-2017 Formulations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC71; U1111-1174-4738 (Other: WHO)
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Influenza; Fluzone® Quadrivalent, Influenza Vaccine (2016-2017 formulation); Fluzone® High-Dose, Influenza Vaccine (2016-2017 formulation)
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years (Experimental): Participants aged 3 to < 9 years received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. For participants for whom 2 doses of influenza vaccine were recommended per Advisory Committee on Immunization Practices (ACIP) guidance, a second dose of Fluzone Quadrivalent vaccine was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, 2016-2017 formulation, No Preservative
- Fluzone Quadrivalent Vaccine Group 2: 18 to < 65 Years (Experimental): Participants aged 18 to < 65 years received one 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0.
  Interventions: Biological: Fluzone Quadrivalent vaccine, 2016-2017 formulation, No Preservative
- Fluzone High-Dose Vaccine Group 3: ≥ 65 Years (Experimental): Participants aged ≥ 65 years received one 0.5-mL dose of Fluzone High-Dose vaccine, intramuscularly, at Day 0.
  Interventions: Biological: Fluzone High-Dose, vaccine, 2016-2017 formulation

INTERVENTIONS:
Biological: Fluzone Quadrivalent vaccine, 2016-2017 formulation, No Preservative — 0.5 mL, Intramuscular
  Other Names: Fluzone® Quadrivalent, Influenza Vaccine
  Arms: Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years
Biological: Fluzone Quadrivalent vaccine, 2016-2017 formulation, No Preservative — 0.5 mL, Intramuscular
  Other Names: Fluzone® Quadrivalent, Influenza Vaccine
  Arms: Fluzone Quadrivalent Vaccine Group 2: 18 to < 65 Years
Biological: Fluzone High-Dose, vaccine, 2016-2017 formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone® High-Dose Influenza Vaccine
  Arms: Fluzone High-Dose Vaccine Group 3: ≥ 65 Years

SUMMARY:
The aim of the study was to describe the safety and immunogenicity of the 2016-2017 formulations of Fluzone Quadrivalent vaccine in children 3 to < 9 years of age and in adults 18 to < 65 years or age, and of the 2016-2017 formulation of Fluzone High-Dose vaccine in adults ≥65 years of age.

Primary Observational Objectives

* To describe the safety of the 2016-2017 formulation of Fluzone Quadrivalent vaccine in children 3 to < 9 years of age and adults 18 to < 65 years of age, and the safety of the 2016-2017 formulation of Fluzone High-Dose vaccine in adults ≥ 65 years of age.

Observational Objectives:

* To describe the immunogenicity of the 2016-2017 formulation of Fluzone Quadrivalent vaccine in children 3 to < 9 years of age and adults 18 to < 65 years of age, and the immunogenicity of the 2016-2017 formulation of Fluzone High-Dose vaccine in adults ≥ 65 years of age.
* To submit available sera from approximately 90 participants (30 participants 3 to < 9 years of age and 30 participants 18 to < 65 years of age who receive Fluzone Quadrivalent vaccine, and 30 participants ≥ 65 years of age who receive Fluzone High-Dose vaccine) to Center for Biologics Evaluation and Research (CBER) for further analysis by the World Health Organization (WHO), the Centers for Disease Control and Prevention (CDC), and the Food and Drug Administration (FDA) to support formulation recommendations for subsequent influenza vaccines.

DETAILED DESCRIPTION:
All participants received a 0.5-mL intramuscular dose of their assigned vaccine at Visit 1. For participants 3 to < 9 years of age for whom 2 doses of influenza vaccine were recommended per Advisory Committee on Immunization Practices (ACIP) guidance, a second dose of Fluzone Quadrivalent vaccine (of the same volume) was administered during Visit 2.

Solicited adverse reaction (AR) information was collected for 7 days after vaccination. Unsolicited non-serious adverse event (AE) and serious adverse event (SAE) information was collected from Visit 1 to Visit 2 or from Visit 1 to Visit 3 for those participants receiving 2 doses of study vaccine.

Immunogenicity was evaluated in all participants prior to vaccination on Day 0 (Visit 1) and after the final vaccination on Day 28 for 3 to < 9 year olds and Day 21 days for adults 18 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 to <9 years or adult aged ≥ 18 years on the day of first study vaccination (study product administration) .
* Informed consent form had been signed and dated by participants ≥ 18 years of age.
* Assent form had been signed and dated by participants 7 to <9 years of age, and informed consent form (ICF) has been signed and dated by parent(s) or guardian(s) for participants 3 to <9 years of age.
* Participant and parent/guardian (of participants 3 to <9 years of age) were able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche, or post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment (or in the 30 days preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 30 days preceding the first trial vaccination, or planned receipt of any vaccine before Visit 2 for participants receiving 1 dose of influenza vaccine or Visit 3 for participants receiving 2 doses of influenza vaccine.
* Previous vaccination against influenza (in the 2016-2017 influenza season) with either the trial vaccine or another vaccine.
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Thrombocytopenia, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of planned vaccination or febrile illness (temperature ≥100.4°F [38.0°C]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study (participants ≥18 years of age) or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study (all participants).
* History of serious adverse reaction to any influenza vaccine.
* Personal history of Guillain-Barré syndrome.
* Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-09-15; Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- United States (2):
  - Bardstown, Kentucky
  - Metairie, Louisiana

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 2 centers in the United States from 15 September 2016 to 28 September 2016.
Pre-assignment Details: A total of 180 participants (60 for each group) were enrolled and vaccinated in the study.
Period: Overall Study
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years | Fluzone Quadrivalent Vaccine Group 2: 18 to < 65 Years | Fluzone High-Dose Vaccine Group 3: ≥ 65 Years
Started | 60 | 60 | 60
Completed | 60 | 60 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years: Participants aged 3 to < 9 years received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. For participants for whom 2 doses of influenza vaccine were recommended per ACIP guidance, a second dose of Fluzone Quadrivalent vaccine was administered at Day 28.
- Total: Total of all reporting groups
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years | Fluzone Quadrivalent Vaccine Group 2: 18 to < 65 Years | Fluzone High-Dose Vaccine Group 3: ≥ 65 Years | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.03 (1.61) | 42.2 (12.9) | 72.6 (6.19) | 40.3 (28.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 42 | 45 | 113
  Male | 34 | 18 | 15 | 67
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site Reactions (Pain, Erythema, and Swelling) and Systemic Reactions (Fever, Headache, Malaise, Myalgia): Group 1 (3 to < 9 Years of Age)
Description: Solicited injection site reactions: Pain (Grade 1: easily tolerated, Grade 2: sufficiently discomforting to interfere with normal behavior or activities, Grade 3: incapacitating, unable to perform usual activities), erythema & swelling (Grade 1: >0 to <25 mm;Grade 2: ≥ 25 to < 50 mm; Grade 3: ≥ 50 mm). Solicited systemic reactions: Fever (Grade 1: ≥ 38.0 degrees Celsius to ≤ 38.4 degrees Celsius, Grade 2: ≥ 38.5 degrees Celsius to ≤ 38.9 degrees Celsius, Grade 3: ≥ 39.0 degrees Celsius), headache, malaise & myalgia (Grade 1: no interference with activity, Grade 2: some interference, Grade 3: significant interference). Number of participants with any solicited injection-site & systemic reactions are reported; number of participants with Grade 3 solicited injection-site & systemic reactions are also reported.
Time Frame: Within 7 days after any vaccination
Population: Analysis was performed using the Safety Analysis Set, which included all participants who received the study vaccine. Number of participants analyzed corresponds to participants with available data for the listed solicited reaction.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years
Number analyzed (Participants) | 60
Participants
  Any Injection site pain: number analyzed (Participants) | 58
  Any Injection site pain | 18
  Grade 3 Injection site pain: number analyzed (Participants) | 58
  Grade 3 Injection site pain | 1
  Any Injection site erythema: number analyzed (Participants) | 58
  Any Injection site erythema | 6
  Grade3 Injection site erythema: number analyzed (Participants) | 58
  Grade3 Injection site erythema | 0
  Any Injection site swelling: number analyzed (Participants) | 58
  Any Injection site swelling | 7
  Grade3 Injection site swelling: number analyzed (Participants) | 58
  Grade3 Injection site swelling | 0
  Any Fever: number analyzed (Participants) | 57
  Any Fever | 3
  Grade 3 Fever: number analyzed (Participants) | 57
  Grade 3 Fever | 1
  Any Headache: number analyzed (Participants) | 57
  Any Headache | 9
  Grade 3 Headache: number analyzed (Participants) | 57
  Grade 3 Headache | 0
  Any Malaise: number analyzed (Participants) | 57
  Any Malaise | 15
  Grade 3 Malaise: number analyzed (Participants) | 57
  Grade 3 Malaise | 1
  Any Myalgia: number analyzed (Participants) | 57
  Any Myalgia | 12
  Grade 3 Myalgia: number analyzed (Participants) | 57
  Grade 3 Myalgia | 0

2. Primary Outcome: Number of Participants Reporting Solicited Injection Site Reactions (Pain, Erythema, and Swelling) and Systemic Reactions (Fever, Headache, Malaise, Myalgia): Group 2 (18 to < 65 Years) and Group 3 (≥ 65 Years)
Description: Solicited injection site reactions: Pain (Grade 1: no interference with activity, Grade 2: some interference, Grade 3: significant; prevents daily activity), erythema & swelling (Grade 1: ≥ 25 to ≤ 50 mm; Grade 2: ≥ 51 to ≤ 100 mm; Grade 3: >100 mm). Solicited systemic reactions: Fever (Grade 1: ≥ 38.0 degrees Celsius to ≤ 38.4 degrees Celsius, Grade 2: ≥ 38.5 degrees Celsius to ≤ 38.9 degrees Celsius, Grade 3: ≥ 39.0 degrees Celsius), headache, malaise & myalgia (Grade 1: no interference with activity, Grade 2: some interference, Grade 3: significant interference). Number of participants with any solicited injection-site & systemic reactions are reported; number of participants with Grade 3 solicited injection-site & systemic reactions are also reported.
Time Frame: Within 7 days after any vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone Quadrivalent Vaccine Group 2: 18 to < 65 Years | Fluzone High-Dose Vaccine Group 3: ≥ 65 Years
Number analyzed (Participants) | 60 | 60
Participants
  Any Injection site pain | 28 | 12
  Grade 3 Injection site pain | 0 | 0
  Any Injection site erythema | 0 | 3
  Grade3 Injection site erythema | 0 | 0
  Any Injection site swelling | 0 | 1
  Grade3 Injection site swelling | 0 | 0
  Any Fever | 0 | 1
  Grade 3 Fever | 0 | 0
  Any Headache | 11 | 8
  Grade 3 Headache | 0 | 0
  Any Malaise | 10 | 4
  Grade 3 Malaise | 0 | 0
  Any Myalgia | 15 | 11
  Grade 3 Myalgia | 0 | 0

3. Secondary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies (Group 1: 3 to < 9 Years)
Description: Anti-influenza antibodies were measured using hemagglutination inhibition (HAI) assay for 4 strains: H1N1, H3N2, Victoria lineage, Yamagata lineage.
Time Frame: Day 0 (pre-vaccination) and 28 days post-final vaccination (post-vaccination)
Population: Analysis was performed using the Per-protocol Analysis Set (PPAS), which included all participants who received study vaccine and had a valid post-vaccination serology result for at least 1 strain.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years
Number analyzed (Participants) | 54
Titers (1/dilutions)
  Pre-Vaccination: A/H1N1 | 273 [177 to 419]
  Pre-Vaccination: A/H3N2 | 167 [106 to 265]
  Pre-Vaccination: B Victoria: number analyzed (Participants) | 53
  Pre-Vaccination: B Victoria | 111 [63.1 to 195]
  Pre-Vaccination: B Yamagata | 170 [103 to 279]
  Post-Vaccination: A/H1N1 | 1232 [961 to 1579]
  Post-Vaccination: A/H3N2 | 2495 [1893 to 3289]
  Post-Vaccination: B Victoria | 1208 [807 to 1809]
  Post-Vaccination: B Yamagata | 1731 [1230 to 2435]

4. Secondary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies (Group 2: 18 to < 65 Years)
Description: as for outcome 3
Time Frame: Day 0 (pre-vaccination) and 21 days post-final vaccination (post-vaccination)
Population: Analysis was performed on PPAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | Fluzone Quadrivalent Vaccine Group 2: 18 to < 65 Years
Number analyzed (Participants) | 60
Titers (1/dilutions)
  Pre-Vaccination: A/H1N1 | 225 [151 to 335]
  Pre-Vaccination: A/H3N2 | 66.1 [45.7 to 95.6]
  Pre-Vaccination: B Victoria | 195 [136 to 278]
  Pre-Vaccination: B Yamagata | 264 [181 to 386]
  Post-Vaccination: A/H1N1 | 779 [584 to 1039]
  Post-Vaccination: A/H3N2 | 752 [562 to 1006]
  Post-Vaccination: B Victoria | 998 [787 to 1267]
  Post-Vaccination: B Yamagata | 1470 [1114 to 1941]

5. Secondary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies (Group 3: ≥ 65 Years)
Description: Anti-influenza antibodies were measured using hemagglutination inhibition (HAI) assay for 3 strains: H1N1, H3N2, Victoria lineage.
Time Frame: Day 0 (pre-vaccination) and 21 days post-final vaccination (post-vaccination)
Population: Analysis was performed on PPAS.
Measure: Median (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | Fluzone High-Dose Vaccine Group 3: ≥ 65 Years
Number analyzed (Participants) | 60
Titers (1/dilutions)
  Pre-Vaccination: A/H1N1 | 77.3 [51.8 to 115]
  Pre-Vaccination: A/H3N2 | 59.6 [39.6 to 89.6]
  Pre-Vaccination: B Victoria | 106 [77.4 to 146]
  Post-Vaccination: A/H1N1 | 347 [249 to 484]
  Post-Vaccination: A/H3N2 | 590 [406 to 858]
  Post-Vaccination: B Victoria | 816 [607 to 1097]

6. Secondary Outcome: Number of Participants With Seroprotection to Influenza Vaccine Antigens (Group 1: 3 to < 9 Years)
Description: Anti-influenza antibodies were measured using HAI assay for 4 strains: H1N1, H3N2, Victoria lineage, Yamagata lineage. Seroprotection was defined as an antibody titer ≥40 (1/dilution [dil]) at pre-vaccination and at post-final vaccination.
Time Frame: Day 0 (pre-vaccination) and 28 days post-final vaccination (post-vaccination)
Population: Analysis was performed on PPAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years
Number analyzed (Participants) | 54
Participants
  Pre-Vaccination: A/H1N1 | 46
  Pre-Vaccination: A/H3N2 | 47
  Pre-Vaccination: B Victoria: number analyzed (Participants) | 53
  Pre-Vaccination: B Victoria | 35
  Pre-Vaccination: B Yamagata | 41
  Post-Vaccination: A/H1N1 | 54
  Post-Vaccination: A/H3N2 | 54
  Post-Vaccination: B Victoria | 52
  Post-Vaccination: B Yamagata | 53

7. Secondary Outcome: Number of Participants With Seroprotection to Influenza Vaccine Antigens (Group 2: 18 to < 65 Years)
Description: Anti-influenza antibodies were measured using HAI assay for 4 strains: H1N1, H3N2, Victoria lineage, Yamagata lineage. Seroprotection was defined as an antibody titer ≥ 40 (1/dilution [dil]) at pre-vaccination and at post-final vaccination.
Time Frame: Day 0 (pre-vaccination) and 21 days post-final vaccination (post-vaccination)
Population: Analysis was performed on PPAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone Quadrivalent Vaccine Group 2: 18 to < 65 Years
Number analyzed (Participants) | 60
Participants
  Pre-Vaccination: A/H1N1 | 53
  Pre-Vaccination: A/H3N2 | 40
  Pre-Vaccination: B Victoria | 52
  Pre-Vaccination: B Yamagata | 56
  Post-Vaccination: A/H1N1 | 60
  Post-Vaccination: A/H3N2 | 60
  Post-Vaccination: B Victoria | 60
  Post-Vaccination: B Yamagata | 60

8. Secondary Outcome: Number of Participants With Seroprotection to Influenza Vaccine Antigens (Group 3: ≥ 65 Years)
Description: Anti-influenza antibodies were measured using HAI assay for 3 strains: H1N1, H3N2, Victoria lineage. Seroprotection was defined as an antibody titer ≥ 40 (1/dilution [dil]) at pre-vaccination and at post-final vaccination.
Time Frame: Day 0 (pre-vaccination) and 21 days post-final vaccination (post-vaccination)
Population: Analysis was performed on PPAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone High-Dose Vaccine Group 3: ≥ 65 Years
Number analyzed (Participants) | 60
Participants
  Pre-Vaccination: A/H1N1 | 41
  Pre-Vaccination: A/H3N2 | 39
  Pre-Vaccination: B Victoria | 51
  Post-Vaccination: A/H1N1 | 56
  Post-Vaccination: A/H3N2 | 58
  Post-Vaccination: B Victoria | 60

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to Day 56 for Group 1; up to Day 21 for Groups 2 and 3.
Description: A solicited reaction is an AE that is prelisted in the electronic Case Report Form (eCRF) and considered to be related to vaccination. A solicited reaction is therefore an adverse drug reaction (ADR) observed and reported under the conditions (nature and time to onset) prelisted (i.e., solicited) in the eCRF.
  An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or time to onset post-vaccination.
Arm/Group | Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years | Fluzone Quadrivalent Vaccine Group 2: 18 to < 65 Years | Fluzone High-Dose Vaccine Group 3: ≥ 65 Years
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/60 | 2/60
Other Adverse Events (participants affected / at risk) | 35/60 | 33/60 | 25/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years (N=60) | Fluzone Quadrivalent Vaccine Group 2: 18 to < 65 Years (N=60) | Fluzone High-Dose Vaccine Group 3: ≥ 65 Years (N=60)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluzone Quadrivalent Vaccine Group 1: 3 to < 9 Years (N=60) | Fluzone Quadrivalent Vaccine Group 2: 18 to < 65 Years (N=60) | Fluzone High-Dose Vaccine Group 3: ≥ 65 Years (N=60)
Injection site erythema (General disorders) | 6 | 0 | 3
Injection site pain (General disorders) | 18 | 28 | 12
Injection site swelling (General disorders) | 7 | 0 | 1
Malaise (General disorders) | 15 | 10 | 4
Pyrexia (General disorders) | 5 | 0 | 1
Bronchiolitis (Infections and infestations) | 3 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 4 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 15 | 12
Headache (Nervous system disorders) | 9 | 11 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.